CLINICAL TRIAL: NCT06586892
Title: Quantitative Imaging Biomarker Prospective Validation of Dynamic Contrast-enhanced MRI as a Metric of Orodental Injury After Radiotherapy (QI-ProVE-MRI)
Acronym: (QI-ProVE-MRI)
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2024-0406; NCI-2024-06902 (Other: National Cancer Institute)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Orodental Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Radiotherapy followed by chemotherapy — Researchers would like to test the accuracy of the MRI data being used for this study. If you agree, you will have 2 additional MRI scans within 2 weeks before Visit 1.
  The first 90 participants who agree will be selected to have the following scans:
  * 35 participants will be scanned 2 times on one MRI device (Device #1).
  * 35 participants will be scanned 2 times on another MRI device (Device #2).
  * 20 participants will be scanned 1 time on both MRI devices (Device #1 and #2). If you agree and you are chosen, the study doctor will tell you if you will have scans on
    1. or 2 MRI devices.

SUMMARY:
This research will focus on the prospective qualification and validation of dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) candidate biomarkers (i.e., Ktrans and Ve) to assess the natural history of osteoradionecrosis (ORN) and treatment for this devastating complication related to irradiation of head and neck cancers. The investigations will also include assessment of DCE-MRI candidate biomarkers for pre-qualification as quantitative imaging biomarkers of soft-tissue structures.

DETAILED DESCRIPTION:
This prospective observational study will acquire DCE-MRI data from 200 evaluable patients, specifically with an elevated dosimetric risk to assure an event rate of 20% by 36 months post-radiation, sufficient to demonstrate biomarker performance in the clinical cohort most reflective of relative ORN risk. The final study cohort will consist of individuals undergoing definitive radiotherapy for primary head and neck malignancy. The study subjects will include patients with primarily elevated risk of ORN based on clinical (e.g., pre-RT dental procedures) and dosimetric risk factors we established in prior work (e.g., D30>50Gy, V44 ≥ 42%, or V58 ≥ 25%). All subjects will receive standard IMRT or IMPT as part of their standard clinical care, and treatment plans delivered will be in no way modified based on experimental imaging. Multi-parametric DCE-MRI imaging will be serially performed as per this study's manual of procedures. Clinical data regarding for evaluation of possible dental, mandibular, as well as other normal tissue organs-at-risk side effects will be collected prospectively from medical and dental records for correlation with the DCE-MRI imaging biomarkers. Functional outcomes and patient-reported outcomes questionnaires will be completed to detail outcomes of the continuum of treatment and survivorship.

ELIGIBILITY:
Inclusion Criteria:

Provide signed and dated informed consent form.

* Aged 18 years or older.
* Have histologic evidence of malignant neoplasm that may have been obtained from the primary tumor or metastatic lymph node.
* Have a clinical decision made to receive external beam radiation therapy (EBRT) with curative intent, with or without concomitant chemotherapy.
* Have a good performance status (ECOG score 0-2) evaluated during screening (4 weeks prior to baseline imaging).
* Be willing to comply with all study procedures.
* Be willing to participate for the duration of the study.
* Have elevated dosimetric risk mainly characterized by any of the following criteria:

  * D30>50Gy: 30% of the whole-mandible volume received a dose greater than 50 Gy
  * V44 ≥ 42%: at least 42% of the volume received a dose of 44 Gy or more or
  * V58 ≥ 25%: at least 25% of the volume received a dose of 58 Gy or more.

Exclusion Criteria:

Unable to tolerate DW-MRI or DCE-MRI;

* Having an estimated GFR < 30 ml/min/1.73 m2;
* Contraindication to MRI (e.g., non-MRI compatible metallic implants)
* Pregnant females
* Unable or unwilling to give written, informed consent to undergo MRI imaging.
* Claustrophobia
* Unable to obtain imaging studies of adequate quality to assess imaging-based biomarkers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lai, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org